CLINICAL TRIAL: NCT06118723
Title: The SUPRAMAX-study: Supramaximal Resection Versus Maximal Resection for High-Grade Glioma Patients (ENCRAM 2201)
Brief Title: The SUPRAMAX Study: Supramaximal Resection Versus Maximal Resection for High-Grade Glioma Patients (ENCRAM 2201)
Acronym: SUPRAMAX
Status: Recruiting | Type: Observational
Sponsor: Jasper Gerritsen (Other)
Collaborators: Haaglanden Medical Centre (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital Heidelberg (Other); Technical University of Munich (Other); Insel Gruppe AG, University Hospital Bern (Other); Massachusetts General Hospital (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Jasper Gerritsen, Dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2020-0812-2
Record Dates: First submitted 2023-10-12; First posted 2023-11-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma; High-grade Glioma; Glioblastoma, IDH-wildtype; Glioblastoma, IDH-mutant; Glioblastoma Multiforme, Adult; Astrocytoma, Grade IV; Astrocytoma, Grade III; Astrocytoma, Malignant; Brain Neoplasms; Brain Neoplasm, Primary; Brain Neoplasms, Adult; Brain Neoplasm, Malignant
Keywords: Glioblastoma; Supramaximal resection; FLAIRectomy; Non-contrast enhancement; Neurological morbidity; Quality of life; Overall survival; Progression-free survival
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supramaximal resection: Supramaximal resection: maximal resection of the contrast-enhancing and non-contrast-enhancing part of the tumor (FLAIRectomy)
  Interventions: Procedure: Supramaximal resection
- Maximal safe resection: Maximal safe resection of the contrast-enhancing part of the tumor
  Interventions: Procedure: Maximal safe resection

INTERVENTIONS:
Procedure: Supramaximal resection — Supramaximal resection. Tumor resection continues until either the FLAIR abnormalities have been resected based on the neuronavigation (after updating the navigation intraoperatively), or when subcortical tracts are identified with intraoperative stimulation.
  Other Names: Supramarginal resection; FLAIRectomy; Resection of the non-contrast-enhancing tumor
  Groups: Supramaximal resection
Procedure: Maximal safe resection — Maximal safe resection. Tumor resection continues until maximal safe resection has been achieved as by the neurosurgeon's opinion.
  Groups: Maximal safe resection

SUMMARY:
A greater extent of resection of the contrast-enhancing (CE) tumor part has been associated with improved outcomes in high-grade glioma patients. Recent results suggest that resection of the non-contrast-enhancing (NCE) part might yield even better survival outcomes (supramaximal resection, SMR). Therefore, this study evaluates the efficacy and safety of SMR with and without mapping techniques in HGG patients in terms of survival, functional, neurological, cognitive, and quality of life outcomes. Furthermore, it evaluates which patients benefit the most from SMR, and how they could be identified preoperatively.

This study is an international, multicenter, prospective, 2-arm cohort study of observational nature. Consecutive HGG patients will be operated with supramaximal resection or maximal resection at a 1:3 ratio. Primary endpoints are: 1) overall survival and 2) proportion of patients with NIHSS (National Institute of Health Stroke Scale) deterioration at 6 weeks, 3 months, and 6 months postoperatively. Secondary endpoints are 1) residual CE and NCE tumor volume on postoperative T1-contrast and FLAIR MRI scans 2) progression-free survival; 3) onco-functional outcome, and 4) quality of life at 6 weeks, 3 months, and 6 months postoperatively.

The study will be carried out by the centers affiliated with the European and North American Consortium and Registry for Intraoperative Mapping (ENCRAM).

DETAILED DESCRIPTION:
This is an international, multicenter, prospective, observational, 2-arm cohort study (registration: clinicaltrials.gov ID number TBA). Eligible patients are operated with supramaximal resection versus maximal resection with a 1:3 ratio with a sequential computer-generated random number as subject ID. Intraoperative mapping techniques and/or surgical adjuncts can be used in both treatment arms to ensure the safety of the resection (to minimize the risk of postoperative deficits). Supramaximal resection is defined as 0 cm3 CE tumor and 5 cm3 or less NCE tumor, whereas maximal resection is defined as 0 cm3 CE tumor and >5 cm3 NCE tumor (in line with the updated RANO criteria).

Study patients are allocated to either the supramaximal or maximal safe resection group and will undergo evaluation at presentation (baseline) and during the follow-up period at 6 weeks, 3 months, and 6 months postoperatively. Motor function will be evaluated using the NIHSS (National Institute of Health Stroke Scale) scale. Language function will be evaluated using a standard neurolinguistic test-battery consisting of the Aphasia Bedside Check (ABC), Shortened Token test, Verbal fluency, Picture description and Object naming. Cognitive function will be assessed using the Montreal Cognitive Assessment (MOCA). Patient functioning with be assessed with the Karnofsky Performance Scale (KPS) and the ASA (American Society of Anesthesiologists) physical status classification system. Health-related quality of life (HRQoL) will be assessed with the EORTC QLQ C30, EORTC QLQ BN20 and EQ 5D questionnaires. Overall survival and progression-free survival will be assessed. We expect to complete patient inclusion in 4 years. The estimated duration of the study (including follow-up) will be 5 years.

The primary study objective is to evaluate the safety and efficacy of supramaximal resection versus safe maximal resection in HGG patients as measured by overall survival (OS) and postoperative NIHSS deterioration. Secondary study objectives are to evaluate extent of resection of CE and NCE tumor, quality of life, progression-free survival (PFS), onco-functional outcome (OFO), and SAEs after SMR or maximal safe resections as measured by volumetric analyses of contrast-enhanced MRI images with gadolinium combined with FLAIR images, tumor progression on MRI scans, quality of life questionnaires (EORTC QLQ C30, EORTC QLQ BN20, EQ 5D), combining postoperative residual volume with NIHSS outcomes, and recording SAEs respectively.

Patients will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Tumor diagnosed as HGG (WHO grade III/IV) on MRI as assessed by the neurosurgeon
3. Written informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brainstem or midline
2. Multifocal contrast enhancing lesions
3. Medical reasons precluding MRI (e.g. pacemaker)
4. Inability to give written informed consent
5. Secondary high-grade glioma due to malignant transformation from low-grade glioma
6. Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary high-grade glioma will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.
Sampling Method: Non-Probability Sample
Enrollment: 784 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years postoperatively
  Time from diagnosis to death from any cause
Neurological morbidity at 6 weeks | 6 weeks postoperatively
  NIHSS deterioration of 1 point or more at 6 weeks after surgery

SECONDARY OUTCOMES:
Neurological morbidity at 3 months | 3 months postoperatively
  NIHSS deterioration of 1 point or more at 3 months after surgery
Neurological morbidity at 6 months | 6 months postoperatively
  NIHSS deterioration of 1 point or more at 6 months after surgery
Progression-free survival | Up to 5 years postoperatively
  Time from diagnosis to disease progression (occurrence of a new tumor lesions with a volume greater than 0.175 cm3, or an increase in residual tumor volume of more than 25%) or death, whichever comes first
Residual tumor volume | Within 72 hours postoperatively
  Residual tumor volume of the contrast-enhancing and non-contrast enhancing part, as assessed by a neuroradiologist on postoperative MRI scan (T1 with contrast and FLAIR sequences) using manual or semi-automatic volumetric analyses (Brainlab Elements iPlan CMF Segmentation, Brainlab AG, Munich, Germany; or similar software)
Onco-functional outcome | 6 weeks postoperatively
  According to the OFO classification, consisting of the combination of presence/absence of functional deterioration with gross-total resection
Quality of life at 6 weeks (EORTC QLQ C30) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 weeks (EORTC QLQ BN20) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 weeks (EQ-5D) | 6 weeks postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 3 months (EORTC QLQ C30) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 3 months (EORTC QLQ BN20) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 3 months (EQ-5D) | 3 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 6 months (EORTC QLQ C30) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 months (EORTC QLQ BN20) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 months (EQ-5D) | 6 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Serious Adverse Events | 6 weeks postoperatively
  Serious Adverse Events within 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Gerritsen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- United States (2):
  - University of California, San Francisco (UCSF), San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Hospitals Leuven, Leuven, Belgium
- Germany (2):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Technical University Munich, Munich, Bavaria
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haaglanden Medical Centre, The Hague, South Holland
- Inselspital Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided